CLINICAL TRIAL: NCT02303249
Title: Interventional Study of Videoconferences Between Hospital and Municipality After Discharge From Roskilde and Køge Hospitals - a Randomized Controlled Trial
Brief Title: Interventional Study of Videoconferences Between Hospital and Municipality - a Randomized Controlled Trial
Acronym: Tele-hjem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Region Zealand (Other); Roskilde Municipality (Unknown); Køge Municipality (Unknown); Stevns Municipality (Unknown); Solrød Municipality (Unknown); Lejre Municipality (Unknown); Faxe Municipality (Unknown); Greve Municipality (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SJ-337
Record Dates: First submitted 2014-11-07; First posted 2014-11-27 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Discharge Planning; Readmission, Hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Review of discharges and cross-sectoral video conferencing immediately after discharge
  Interventions: Other: Review of discharges and cross-sectoral video conferencing immediately after discharge
- Control (No Intervention): Standard health care services

INTERVENTIONS:
Other: Review of discharges and cross-sectoral video conferencing immediately after discharge — The intervention is video conference which is randomized and is an intervention that is assigned by the investigator.
  Arms: Intervention

SUMMARY:
The study aims to assess whether the review of discharge planning followed by a cross-sectoral video conference in connection with discharge of medical and geriatric patients at Roskilde and Køge hospitals as well as patients from the Emergency Department at Køge Hospital reduces the proportion of patients who are readmitted within 180 days.

Project nurses at the two hospitals identifies all patients fulfilling the inclusion criteria (above 55 years of age, discharged to their own home), get informed consent and performs the video conferences. Within a few hours after discharge a video conference is held in the patient´s home including the patient,the municipal nurse and the project nurse at the hospital. During the video conference the discharge is reviewed using a structured assessment.

The survey is conducted as an open, randomized intervention study.

DETAILED DESCRIPTION:
The study consists of two parts: First, the project nurse reviews the patients discharge together with the nurse from the hospital ward. Next, the patient is discharged from the hospital and meets the nurse from the municipality at home. Together with the patient the nurse form the municipality reviews:

* Documents from the hospital
* Medicine
* Nutrition
* Mobility
* Assessment of the need for health care services from the municipality

All patients in the project - both patients in the intervention group and patients in the control group - will receive treatment and care equivalent to normally applicable quality standards.

In 2011 4387 patients were discharged Monday to Friday from the Medical and Geriatric Departments at Roskilde and Køge Hospital to one of the seven municipalities. Of these, 1204 persons (27%) were readmitted (in any department) within 180 days. It is expected that the study demonstrates a reduction of ≥ 6 percentage points (from 27% to 21%) with a power of 80% and a significance level of 5%. There will be a need for 792 patients in both control and intervention group, ie 1584 in total.

ELIGIBILITY:
Inclusion Criteria:

* Discharge from the Medical Department and Geriatric Department at Roskilde and Køge hospitals or the Emergency Department at Køge Hospital.

Address in Køge, Greve, Faxe, Solrød, Lejre, Stevns or Roskilde municipalities. Discharges between 8 am and 4 pm Monday-Friday. Acute/subacute admission to the hospital

Exclusion Criteria:

* Patients who cannot give consent to participation. Discharge to a nursing home or relief care home. Patients with planned readmission. Former participant in the study. Patients who are included in the Sub Acute Project. Patients who needs terminal care

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1387 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who are readmitted | 180 days
  Acute readmissions to any hospital in Denmark

SECONDARY OUTCOMES:
Use of municipal services (nursing, practical help, personal care) | 4 months
Time to readmission | 180 days
Total number of readmissions | 180 days
Total number of days of readmission | 180 days
The number of contacts with general practitioner | 180 days
Death | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Solvejg Henneberg Pedersen, dr., Study Director — Region Zealand; Birgitte Dreyer Sørensen, cand. scient. san. publ., Principal Investigator — Region Zealand
Locations (1):
- Region Zealand, Roskilde and Køge Hospitals, Køge, Denmark